CLINICAL TRIAL: NCT06225973
Title: A Phase 2b, Multicenter, Randomized, Double-masked Vehicle-controlled Study to Evaluate the Efficacy and Safety of TL-925 Ophthalmic Emulsion 0.1% in Subjects With Moderate to Severe Dry Eye Disease
Brief Title: A Study of TL-925 Ophthalmic Emulsion as a Treatment for Dry Eye Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TL-925-303
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sponsor, Investigators and study staff will be masked during the randomization process and throughout the study. The study site will have the capacity to unmask participants in an emergency.
  Following completion of the study, the randomization code will be unmasked once all data has been entered into the study database for every subject and the database has been locked.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TL-925 Arm (Experimental): TL-925 will be administered OU BID
  Interventions: Drug: TL-925
- Vehicle Arm (Placebo Comparator): Vehicle will be administered OU BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TL-925 — TL-925 is an eye drop.
  Arms: TL-925 Arm
Other: Placebo — The composition of the vehicle is identical to the active formulation except for the exclusion of the active ingredient.
  Arms: Vehicle Arm

SUMMARY:
In this prospective, phase 2b, multicenter, randomized, double-masked, vehicle-controlled, parallel-arm study, approximately 880 subjects with moderate to severe dry eye disease (DED) will be randomly assigned (1:1) to receive either TL-925 or vehicle as topical ophthalmic eye drops administered bilaterally BID.

The study will comprise two phases: a two-week screening phase/run-in and a six-week double-masked treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dry eye disease for at least 6 months
* An unanesthetized Schirmer's test score (STS) of ≤ 10mm and ≥ 1mm in the study eye
* Female subjects of childbearing potential and their male partners must both use a highly effective contraception method during the study

Exclusion Criteria:

* Any clinically significant slit lamp finding
* Any ongoing ocular infection (bacterial, viral or fungal) or active ocular inflammation
* Best-corrected visual acuity ≥0.7 logarithm of the minimum angle of resolution
* Any keratorefractive surgery within the last 12 months
* Any intraocular or extraocular surgery within 3 months
* Any blepharoplasty or corneal transplant in either eye
* Any form of punctual, or intracanalicular occlusion in either eye
* History or presence of any ocular disorder that may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of TL-925 compared to vehicle on tear production | Baseline to Day 29
  Percentage of subjects who achieve ≥10 mm improvement in Schirmer's test score

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - Nvision - La Mesa, La Mesa, California
  - Nvision - Torrance, Torrance, California
  - Wyse Eyecare, Northbrook, Illinois
  - Pankratz Eye, Columbus, Indiana
  - Butchertown Clinical, Louisville, Kentucky
  - Andover Eye Associates - Andover, Andover, Massachusetts
  - Andover Eye Associates - Raynham, Raynham, Massachusetts
  - NEERA - Westborough, Westborough, Massachusetts
  - NEERA - Woburn, Woburn, Massachusetts
  - Oculus Research, Garner, North Carolina
  - Wilmington Eye, Leland, North Carolina
  - Scott and Christie EyeCare Associates, Cranberry Township, Pennsylvania
  - Advancing Vision Research, Goodlettsville, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, Smyrna, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia